CLINICAL TRIAL: NCT06010277
Title: The Effect of Oral Folinic Acid Rescue Therapy on Pemetrexed Induced Neutropenia: A Randomized Open-label Trial
Brief Title: Folinic Acid for Prevention of Pemetrexed-induced Toxicity
Acronym: FLEX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amphia Hospital (Other)
Collaborators: Albert Schweitzer Hospital (Other)
Responsible Party: Principal Investigator, Dr. N. (Nikki) de Rouw, Dr. Nikki de Rouw, principal investigator, Amphia Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1891
Record Dates: First submitted 2023-01-26; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: NSCLC; Mesothelioma; Thymoma
MeSH Terms: conditions — Mesothelioma; Thymoma | interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folinic acid arm (Experimental): Patients in the intervention-arm will receive oral folinic acid orally 4 times 45mg / day for 3 days, starting 24 hours after the administration of pemetrexed.
  Interventions: Drug: Folinic acid
- No folinic acid arm (No Intervention): Patients will be treated according to regular care.

INTERVENTIONS:
Drug: Folinic acid — Follow-up will take place during the first 4 cycles of chemotherapy with pemetrexed. Patients in the intervention-arm will receive oral folinic acid orally 4 times 45mg / day for 3 days, starting 24 hours after the administration of pemetrexed.
  Arms: Folinic acid arm

SUMMARY:
Objective The main objective is to evaluate the haematological toxicity in patients who use pemetrexed with and without rescue therapy with folinic acid.

Primary endpoint Difference between treatment groups in neutrophil count (*109/L) at day 8-10 after administration of pemetrexed (nadir).

Secondary endpoints The grade neutropenia (according to the CTCAE version 5, 2017) at day 8-10, the homocysteine plasma levels at baseline (predictor for developing toxicity), the efficacy of chemotherapy treatment based on response CT after cycle 2 and 4 and the incidence of discontinuation, dose delays and dose reductions of pemetrexed.

Trial design The FLEX-trial is a multi-centre, open label, double arm, randomized trial to compare neutropenia in patients with and without folinic acid rescue therapy where subjects are participating for 4 treatment cycles.

Population In total 50 patients (25 in each arm), >18 years with stage IV non-small cell lung cancer (NSCLC) or mesothelioma treated with pemetrexed (in combination with other chemo- or immunotherapy) are eligible for inclusion.

Interventions Follow-up will take place during the first 4 cycles of chemotherapy with pemetrexed. Patients in the intervention-arm will receive oral folinic acid orally 4 times 45mg / day for 3 days, starting 24 hours after the administration of pemetrexed.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. ≥18 years old
2. Eligible for treatment with pemetrexed-based chemotherapy based on indication.
3. ECOG performance score of 0-2.
4. Subject is able and willing to sign the Informed Consent Form

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Contraindications for treatment with folinic acid in line with the SmPC.

   1. Hypersensitivity to the active substance or to any of the excipients.
   2. Anaemia caused by vitamin B12 deficiency.
2. The presence of clinically relevant drug-drug interactions, according to the current SmPC of folinic acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Difference in neutrophil count (*109/L) at day 8-10 after pemetrexed administration during 2 cycles of chemotherapy | Between day 8-10 in the first 2 cycles (each cycle is 21 days)
  To evaluate the haematological toxicity (continuous measure) in patients who use pemetrexed with and without rescue therapy with folinic acid.

SECONDARY OUTCOMES:
Grade neutropenia (according to the CTCAE version 5, 2017) at day 8-10 after pemetrexed administration during 2 cycles of chemotherapy | Between day 8-10 in the first 2 cycles (each cycle is 21 days)
  To evaluate the difference in haematological toxicity based on the CTCAE criteria for neutrophil count
Homocysteine plasma levels at baseline (μmol/L) | Once, before the start of the first cycle (each cycle is 21 days)
  To evaluate the influence of baseline homocysteine plasma levels on occurrence of haematological toxicity.
Efficacy based on response CT after cycle 2 and 4 (categorical: response, partial response, progression) | After the second and fourth cycle (each cycle is 21 days)
  To evaluate the efficacy of the treatment with pemetrexed (based on CT-scan).
Incidence of discontinuation, dose delays and dose reductions of pemetrexed | 3 months
  To evaluate the incidence of treatment delay or dose reduction of pemetrexed.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amphia Hospital, Breda, North Brabant
  - Albert Schweitzer Hospital, Dordrecht, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT06010277/Prot_SAP_000.pdf